CLINICAL TRIAL: NCT05570617
Title: The TRACE Study: TRansition to Adulthood Through Coaching and Empowerment - A Pilot Randomized-Controlled Trial
Brief Title: Transition to Adulthood Through Coaching and Empowerment
Acronym: TRACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TRACE
Record Dates: First submitted 2022-09-15; First posted 2022-10-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-11

CONDITIONS: Juvenile Idiopathic Arthritis; Inflammatory Bowel Diseases
Keywords: Transition in care; Empower Youth in their Transition to Adulthood
MeSH Terms: conditions — Arthritis, Juvenile; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition Coach Intervention (Experimental): Half (53) of the participants will be randomly allocated to the Transition Coach Intervention arm of the study. Individuals in the Transition Coach Intervention group will receive the current standard of care (receiving the Youth Transition Roadmap) and meet with the transition coach six times and with a clinical psychologist two times over the course of six months. The meetings between the participant and TC/psychologist will occur over the phone or using the Ontario Telemedicine Network or EPIC.
  Interventions: Behavioral: Transition Coach Intervention
- Standard of Care (Active Comparator): The other half of participants will only receive the current standard of care is the Youth Transition Roadmap which has been developed by Hamilton Health Sciences and provides patients information about 5 domains of healthcare transition; Self-Advocacy, Medication Management, General Health, Lifestyle Issues and Future Planning related to education and vocation.
  Interventions: Behavioral: Standard of Care- Youth Transition Roadmap

INTERVENTIONS:
Behavioral: Transition Coach Intervention — The Transition Coach Intervention will include 8, 1-hour sessions over 6-months. The transition coach will independently meet one-on-one with each youth using an individualized, patient-centred approach beginning with an introductory session, followed by 5 sessions covering each topic in the Youth Transition Roadmap. These topics include: Self-Advocacy, Medication Management, General Health, Lifestyle Issues and Future Planning related to education and vocation. The clinical psychologist will lead 2 sessions beginning with the Patient Health Questionnaire for Anxiety and Depression as a screening tool. The clinical psychologist will discuss psychological and social well-being in the context of their disease covering personally relevant issues/concerns.
  Arms: Transition Coach Intervention
Behavioral: Standard of Care- Youth Transition Roadmap — All participants will receive the Youth Transition Roadmap (standard of care) which discusses 5 domains of healthcare transition; Self-Advocacy, Medication Management, General Health, Lifestyle Issues and Future Planning related to education and vocation. This is an informational pamphlet and will not require any additional meetings with the patient beyond their normal healthcare interactions
  Arms: Standard of Care

SUMMARY:
Pediatric patients with Juvenile Idiopathic Arthritis or Inflammatory Bowel Disease who are preparing to transition into adult care face many unique challenges, and, to date, there is no comprehensive and implementable model of transition care in Canada or the United States. These patients, in addition to the systemic inflammatory nature of their diseases, are also in a period of immense psycho-social stress due to changes in school structure, employment, and general psycho-social growth. A poorly managed transition can have adverse effects on the quality and experience of care as well as contribute to poor disease outcomes including increased morbidity and even mortality.

The goal of this study is to determine the feasibility of using a transition coach intervention to help patients in their transition from pediatric to adult care.

DETAILED DESCRIPTION:
This pilot, feasibility study aims to investigate a new approach to transition from pediatric to adult healthcare for Juvenile Idiopathic Arthritis or Inflammatory Bowel Disease patients.

The study population that will be recruited are 16-17-year-olds with Juvenile Idiopathic Arthritis or Inflammatory Bowel Disease seen in pediatric rheumatology or Gastroenterology clinics.

Upon consent, the patients will be asked by the study coordinator about their preferred method of communication (email or phone). Participants will then be randomly allocated to the Transition Coach Intervention or the control group (standard of care) using the Robust Randomization App using variable permuted block randomization (4 or 6) and a 1:1 allocation ratio. All participants will receive the Youth Transition Roadmap (standard of care) which discusses 5 domains of healthcare transition; Self-Advocacy, Medication Management, General Health, Lifestyle Issues and Future Planning related to education and vocation. The study coordinator will then invite the patients to complete a baseline study questionnaire on the online REDCap secure platform. This baseline questionnaire will gather information to describe our study population including: age, sex, disease type, age at diagnosis, family history, comorbidities and education stream. The investigators will also collect information regarding 'attitude towards transition' and 'feeling ready' for transition using questionnaire.

Once the patient has given informed consent and baseline demographic data has been collected, patients will be asked to complete the following questionnaires using REDCap: i) PedsQL™ 4.0 Generic Scale (18-25 year-old) to measure physical, emotional, social, and school functioning; ii) Patient Global Assessment, a measure of disease activity; and iii) Patient-Reported Outcomes Measurement Information System (PROMIS®) Self-Efficacy outcomes for Chronic Disease including Self-Efficacy for Managing Daily Activities v1.0, Emotions v1.0, Managing Medications and Treatments v1.0, Social Interactions v1.0, Symptoms v1.0, and Informational Support v2.0.

Individuals in the Transition Coach Intervention group will meet with the transition coach six times and with a clinical psychologist two times over the course of six months. The Transition Coach Intervention will include 8, 1-hour sessions over 6-months. The transition coach will independently meet one-on-one with each youth using an individualized, patient-centred approach beginning with an introductory session, followed by 5 sessions covering each topic in the Youth Transition Roadmap.

Upon completing the Transition Coach Intervention, two groups of 4-6 participants each will be randomly selected to participate in an Emotional Mapping exercise to share their experiences/satisfaction with the Transition Coach Intervention. Quality Improvement methods will be employed by Hamilton Health Science's Patient Experience office to yield an Emotional Map to inform modifications to the intervention for a future study

ELIGIBILITY:
Inclusion Criteria:

* 16-17-year-old Juvenile Idiopathic Arthritis or Inflammatory Bowel Disease patients
* can communicate in English
* have access to a phone (or other communication technology such as a laptop),
* are available over the 9-month follow-up period

Exclusion Criteria:

- cannot communicate in English

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility criteria of pilot study assessed through percent enrolment and completion of program | 9 months
  To determine the proportion of study participants who will attend at least 6 of 8 (80%) sessions of the Transition Coach Intervention aimed at improving self-efficacy and self-management skills. To determine the number of patients that cannot consent because of the English language barrier, speech, language, hearing, or visual disability barriers, or technology barrier. To determine the number of patients who consent from the total eligible patients approached. To determine the number of outcome assessments completely and how many data items are missing from the data collection forms. Finally, to determine the number of participants which are satisfied with the number of appointments and timeline of the Transition Coach Intervention.

SECONDARY OUTCOMES:
Preliminary effect of Transition Coach Intervention on changes in self-efficacy as assessed by PROMIS questionnaire for Managing Chronic Conditions- Managing Emotions | 9 months
  Descriptive statistics will summarize patient characteristics and clinical outcomes at each time point. The investigators will describe within-person, within-group and between-group changes in PROMIS® outcomes in both groups using means and standard deviations or medians and interquartile ranges as appropriate.
Preliminary effect of Transition Coach Intervention on changes in self-efficacy as assessed by PROMIS questionnaire for Managing Chronic Conditions- Managing Medications | 9 months
  Descriptive statistics will summarize patient characteristics and clinical outcomes at each time point. The investigators will describe within-person, within-group and between-group changes in PROMIS® outcomes in both groups using means and standard deviations or medians and interquartile ranges as appropriate.
Preliminary effect of Transition Coach Intervention on changes in self-efficacy as assessed by PROMIS questionnaire for Managing Chronic Conditions- Managing Social Interactions | 9 months
  Descriptive statistics will summarize patient characteristics and clinical outcomes at each time point. The investigators will describe within-person, within-group and between-group changes in PROMIS® outcomes in both groups using means and standard deviations or medians and interquartile ranges as appropriate.
Preliminary effect of Transition Coach Intervention on changes in self-efficacy as assessed by PROMIS questionnaire for Managing Chronic Conditions- Managing Symptoms | 9 months
  Descriptive statistics will summarize patient characteristics and clinical outcomes at each time point. The investigators will describe within-person, within-group and between-group changes in PROMIS® outcomes in both groups using means and standard deviations or medians and interquartile ranges as appropriate.
Preliminary effect of Transition Coach Intervention on changes in self-efficacy as assessed by PROMIS questionnaire for Managing Chronic Conditions- Managing Daily Activities | 9 months
  Descriptive statistics will summarize patient characteristics and clinical outcomes at each time point. The investigators will describe within-person, within-group and between-group changes in PROMIS® outcomes in both groups using means and standard deviations or medians and interquartile ranges as appropriate.
Preliminary effect of Transition Coach Intervention on changes in self-efficacy as assessed by PROMIS questionnaire for Informational Support | 9 months
  Descriptive statistics will summarize patient characteristics and clinical outcomes at each time point. The investigators will describe within-person, within-group and between-group changes in PROMIS® outcomes in both groups using means and standard deviations or medians and interquartile ranges as appropriate.
Understand the perspective and experience of youth about the Transition Coach Intervention with a satisfaction questionnaire | 9 months
  Measuring all the participants satisfaction with the Transition Coach Intervention by asking participants to fill in a satisfaction questionnaire asking about the appropriate number of meetings, length of meetings, and the types of topics discussed. The investigators will describe within-person, within-group and between-group changes in satisfaction in both groups using means and standard deviations or medians and interquartile ranges as appropriate.
Understand the perspective and experience of youth about the Transition Coach Intervention with a focus group | 9 months
  Measuring the participants satisfaction with the Transition Coach Intervention by asking participants to join a focus group to do an Emotional Mapping feedback exercise. This will be done by two groups of 5-7 participants (one group of Juvenile Idiopathic Arthritis patients and another of Inflammatory Bowel Disease patients), randomly selected to share their experiences/satisfaction with the Transition Coach Intervention. The responses from the Emotional Mapping exercise will inform modifications to the intervention in the future study.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391